CLINICAL TRIAL: NCT03416010
Title: Healthy Lifestyle Intervention for High-Risk Minority Pregnant Women: A-RCT
Brief Title: Healthy Lifestyle Intervention for High-Risk Minority Pregnant Women
Acronym: A-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); New York University (Other); Jacobi Medical Center (Other); Boston College (Other); University of Arizona (Other); Drexel University (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH); University of South Florida (Other)
Responsible Party: Principal Investigator, Bernadette Melnyk, Dean and Professor, College of Nursing Vice President of Health Promotion, Professor of Pediatrics and Psychiatry, College of Medicine, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2017B0425; 1R01MD012770-01A1 (NIH)
Record Dates: First submitted 2017-11-14; First posted 2018-01-30 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Emotional Disturbances; Depression; Pregnancy Late; Post-Partum Depression; Anxiety; Nutritional Deficiency
Keywords: emotional distress pregnancy disparities minority depression
MeSH Terms: conditions — Affective Symptoms; Depression; Depression, Postpartum; Anxiety Disorders; Malnutrition

STUDY DESIGN:
Intervention Model Description: longitudinal, randomized block RCT with repeated measures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): In addition to standard prenatal care the PregnancyPlus attention control group for 6 weeks will receive 1.5 hours of ACOG-designed patient education pamphlets. Material will include prenatal and post-partum education.. Dr. Gennaro will conduct the training of the attention control group midwives. The same protocol for assessing fidelity for COPE-P also will be used for assessing fidelity to the attention control intervention
- Intervention (Active Comparator): In addition to standard prenatal care the COPE-P intervention group will also receive 1.5 hours each week for 6 weeks the cognitive-behavior skills building program driven by CBT as the theoretical framework by health care providers trained in COPE-P by Dr. Melnyk. The content of the COPE program is driven by the literature review, the theoretical framework, previous studies of COPE interventions with mothers of preterm infants and prior work with pregnant minority women by our team.
  Interventions: Behavioral: COPE-P

INTERVENTIONS:
Behavioral: COPE-P — Session 1 ABCs (A=Antecedent or Activator event, B=Belief that follows the event, C=Consequence: how you feel and how you behave).
  Session 2 self-esteem and positive self-talk, including ways to build self-esteem and the group provides examples of how to change unhealthy habits into healthy ones.
  Session 3 stress/coping during pregnancy. Physical and emotional responses to stress are discussed along with healthy snacking and healthy ways to cope with typical stresses.
  Session 4 planning, goal setting and the 4-step problem solving process. Session 5 dealing with emotions in healthy ways through positive thinking and effective communication.
  Session 6 coping with stressful situations encountered during pregnancy while continuing to reinforce the thinking-feeling-behaving triangle.
  Arms: Intervention

SUMMARY:
The overall purpose of this application is to evaluate the efficacy of an intervention designed to decrease health disparities in pregnant, emotionally distressed, minority women. This randomized controlled trial will test a six session (spaced over 18 weeks) cognitive behavioral skills building (CBSB) prenatal care intervention (specifically designed and based on prior research for pregnant minority women experiencing emotional distress) at three sites (Jacobi Medical Center, New York City and The Ohio State University Total Health and Wellness Clinic, and The Ohio State University Wexner Medical Center OB/GYN Columbus, Ohio.

DETAILED DESCRIPTION:
A randomized controlled trial will test a cognitive behavioral skills building intervention (COPE-P) in Black and Hispanic women experiencing emotional distress in two sites (New York and Ohio) to determine if the intervention leads to better health behaviors, better psychosocial health (anxiety, stress, and depressive symptoms), and improved birth and post-natal outcomes in women experiencing emotional distress. Developing scalable prenatal interventions designed to improve birth outcomes as well as maternal physical and psychosocial health is essential to decrease health disparities in pregnant minority women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages of 18-40 years old
* Pregnant women experiencing an uncomplicated singleton pregnancy of less than 19 weeks
* Self-identified as either Black or Hispanic
* Able to read and speak English.
* The child participants born to the participants will have their record accessed for data collection.

Exclusion Criteria:

* Women with chronic medical conditions (e.g., hypertension, or diabetes), are currently receiving treatment or therapy for a psychiatric diagnosis, or have participated in this study with a prior pregnancy.
* Women with obstetrical complications, such as preeclampsia, gestational diabetes, or fetal abnormalities.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnancy is only experienced by women so only women are included as study participants.
Enrollment: 299 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette Melnyk, PhD, Principal Investigator — Ohio State University
Locations (3):
- United States (3):
  - Jacobi Medical Center, The Bronx, New York
  - OSU Total Health and Wellness, Columbus, Ohio
  - OSUWMC OB/GYN Clinic, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gennaro S, Melnyk BM, Szalacha LA, Gibeau AM, Hoying J, O'Connor CM, Cooper AR, Aviles MM. Effects of Two Group Prenatal Care Interventions on Mental Health: An RCT. Am J Prev Med. 2024 May;66(5):797-808. doi: 10.1016/j.amepre.2024.01.005. Epub 2024 Feb 5. PMID 38323949

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant recruitment was initiated March 5, 2018, at two medical clinic sites in urban clinics in two states. A third medical clinic site was added to support recruitment in 2019. Recruitment closed April 11, 2022.
Pre-assignment Details: 8,335 participant records were prescreened for eligibility. 6,842 did not meet inclusion criteria. 771 declined to participate. 423 participants consented to participate in the study but were ineligible after completing screening questionnaires (GAD-7, PSS, and EPDS).
Groups:
- Control: In addition to standard prenatal care the PregnancyPlus attention control group for 6 weeks will receive 1.5 hours of ACOG-designed patient education pamphlets. Material will include prenatal and post-partum education. Dr. Gennaro will conduct the training of the attention control group midwives. The same protocol for assessing fidelity for COPE-P also will be used for assessing fidelity to the attention control intervention.
- Intervention: In addition to standard prenatal care the COPE-P intervention group will also receive 1.5 hours each week for 6 weeks the cognitive-behavior skills building program driven by CBT as the theoretical framework by health care providers trained in COPE-P by Dr. Melnyk. The content of the COPE program is driven by the literature review, the theoretical framework, previous studies of COPE interventions with mothers of preterm infants and prior work with pregnant minority women by our team.
  COPE-P: Session 1 ABCs (A=Antecedent or Activator event, B=Belief that follows the event, C=Consequence: how you feel and how you behave).
  Session 2 self-esteem and positive self-talk, including ways to build self-esteem and the group provides examples of how to change unhealthy habits into healthy ones.
  Session 3 stress/coping during pregnancy. Physical and emotional responses to stress are discussed along with healthy snacking and healthy ways to cope with typical stresses.
  Session 4 planning, goal setting and the 4-step problem solving process. Session 5 dealing with emotions in healthy ways through positive thinking and effective communication.
  Session 6 coping with stressful situations encountered during pregnancy while continuing to reinforce the thinking-feeling-behaving triangle.
Period: Timepoint 0 (<19 Weeks Gestation)
Arm/Group | Control | Intervention
Started | 122 | 177
Completed | 111 | 145
Not Completed | 11 | 32
Not completed — medically excluded or aged out prior to initiating intervention | 11 | 32
Period: Timepoint 1 (31 Gestational Weeks)
Arm/Group | Control | Intervention
Started | 111 | 145
Completed | 73 | 95
Not Completed | 38 | 50
Not completed — Withdrawal by Subject | 27 | 38
Not completed — Lost to Follow-up | 11 | 12
Period: Timepoint 2 (6 Weeks Postpartum)
Arm/Group | Control | Intervention
Started | 73 | 95
Completed | 71 | 92
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 3
Period: Timepoint 3 (6 Months Postpartum)
Arm/Group | Control | Intervention
Started | 71 | 92
Completed | 68 | 86
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 1 | 3
Not completed — Missing Data | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 122 | 177 | 299
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 122 | 177 | 299
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (5.3) | 26.4 (5.3) | 26.3 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 177 | 299
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56 | 68 | 124
  Not Hispanic or Latino | 49 | 91 | 140
  Unknown or Not Reported | 17 | 18 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 76 | 118 | 194
  White | 6 | 15 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 40 | 44 | 84
Region of Enrollment [Number; unit: participants]
  United States | 122 | 177 | 299
Enrolled in School [Count of Participants; unit: Participants]
  Enrolled | 103 | 35 | 138
  Not Enrolled | 18 | 140 | 158
  Did not respond | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-reported Healthy Lifestyle Beliefs Timepoint 0 to Timepoint 3
Description: Healthy Lifestyle Beliefs Scale survey will be administered at each of the in-person meetings. This scale taps beliefs about various facets of maintaining a healthy lifestyle. This 16-item is scored on a five point Likert-type scale that ranging from 1 strongly disagree to 5 strongly agree. The minimum score is 16 and the maximum score is 80. The higher the score the higher the beliefs of maintaining a healthy lifestyle.
Time Frame: Timepoint 0 (<19 weeks gestation) to Timepoint 3 (6 month well child visit)
Population: All participants who completed data collection at respective timepoints.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 122 | 177
units on a scale
  Timepoint 0 | 59.044 (0.736) | 59.349 (0.615)
  Timepoint 1: number analyzed (Participants) | 73 | 95
  Timepoint 1 | 64.972 (0.823) | 64.234 (0.720)
  Timepoint 2: number analyzed (Participants) | 71 | 92
  Timepoint 2 | 63.683 (0.880) | 64.614 (0.744)
  Timepoint 3: number analyzed (Participants) | 68 | 86
  Timepoint 3 | 63.328 (0.853) | 63.852 (0.744)
Statistical Analysis 1: Comparison: Control vs Intervention; Null Hypothesis: There was no significant difference in Health Beliefs across those 4 time points; Test type: Other; p < 0.001, two-way ANOVA
Statistical Analysis 2: Comparison: Control vs Intervention; Null hypothesis: There was no significant difference between the full intervention group, COPE-P, and the attention-control group, Preg+, in Health Beliefs, as measured by the Healthy Lifestyle Beliefs measure, at T0 baseline, as well as at time points 1, immediately following the intervention, 2, 6 weeks after the infants' birth, and 3, 6 months after the infants' birth; Test type: Other; p < 0.001, two-way ANOVA
Statistical Analysis 3: Comparison: Control vs Intervention; Null hypothesis: There was no statistically significant interaction between the intervention group and time; Test type: Other; p = 0.009, two-way ANOVA

2. Primary Outcome: Change in Self-reported Anxiety Level From Timepoint 0 to Timepoint 3
Description: The Generalized Anxiety Scale (GAD-7) is a 7-item survey which measures anxiety will be administered at each of the in-person meetings. The GAD-7 is a 7-item, 4-point Likert-type scale ranging from (0) Not at all to (3). Scores range from 0 to 21, with higher scores indicating greater functional impairment related to the patient's experience of anxiety. A score greater than or equal to 10 indicates moderate and higher anxiety and will be used in this study,
Time Frame: Timepoint 0 (<19 weeks gestation) to Timepoint 3 (6 month well child visit)
Population: All participants who completed respective timepoints.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 122 | 177
units on a scale
  Timepoint 0 | 8.647 (0.507) | 9.018 (0.329)
  Timepoint 1: number analyzed (Participants) | 73 | 95
  Timepoint 1 | 5.500 (0.507) | 5.447 (0.444)
  Timepoint 2: number analyzed (Participants) | 71 | 92
  Timepoint 2 | 3.358 (0.526) | 4.114 (0.459)
  Timepoint 3: number analyzed (Participants) | 68 | 86
  Timepoint 3 | 3.853 (0.522) | 4.398 (0.459)
Statistical Analysis 1: Comparison: Control vs Intervention; Null hypothesis: there was no significant difference in anxiety across the 4 time points; Test type: Other; p < 0.001, two-way ANOVA — Threshold for significance: p <0.01
Statistical Analysis 2: Comparison: Control vs Intervention; Null hypothesis: There was no significant difference between the two groups in anxiety at T0 baseline, as well as at timepoint 1(immediately following the intervention), timepoint 2 (6 weeks after the infants' birth), and timepoint 3 (6 months after the infants' birth); Test type: Other; p < 0.001, two-way ANOVA
Statistical Analysis 3: Comparison: Control vs Intervention; Null hypothesis: There was no statistically significant interaction between the intervention group and time; Test type: Other; p < 0.001, two-way ANOVA

3. Primary Outcome: Change in Self-reported Healthy Lifestyle Behaviors From Timepoint 0 to Timepoint 3
Description: The Healthy Lifestyle Behaviors Scale survey will be administered at each of the in-person meetings. Participants respond to each of the 15 items (e.g., I exercised regularly; I talked about my worries) on a 5-point Likert-type scale that ranges from 1 strongly disagree to 5 strongly agree. The minimum score is 15 and the maximum score is 75. The higher the score the higher the healthy lifestyle behaviors are practiced.
Time Frame: Timepoint 0 (<19 weeks gestation) to Timepoint 3 (6 month well child visit)
Population: All participants who completed data collection at respective timepoints.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 122 | 177
units on a scale
  Timepoint 0 | 49.506 (0.903) | 50.669 (0.730)
  Timepoint 1: number analyzed (Participants) | 73 | 95
  Timepoint 1 | 56.194 (0.981) | 56.783 (0.868)
  Timepoint 2: number analyzed (Participants) | 71 | 92
  Timepoint 2 | 53.677 (1.032) | 57.267 (0.897)
  Timepoint 3: number analyzed (Participants) | 68 | 86
  Timepoint 3 | 55.692 (1.032) | 56.209 (0.897)
Statistical Analysis 1: Comparison: Control vs Intervention; Null hypothesis: There was no significant difference in health behaviors across those 4 time points; Test type: Other; p < 0.001, two-way ANOVA
Statistical Analysis 2: Comparison: Control vs Intervention; Test type: Other; p < 0.001, two-way ANOVA
Statistical Analysis 3: Comparison: Control vs Intervention; Null Hypothesis: There was no statistically significant interaction between the intervention group and time; Test type: Other; p < 0.001, two-way ANOVA

4. Primary Outcome: Change in Self-reported Depressive Symptoms From Timepoint 0 to Timepoint 3
Description: The Edinburgh Postnatal Depression Scale (EPDS) is a scale measuring depressive symptoms will be administered at each of the in-person meetings. The Edinburgh Postnatal Depression Scale is a 10 item self-report perinatal depression questionnaire. The scale asks participants to describe how they have felt in the previous week. Unlike other depression screening tools, the EPDS excludes questions regarding somatic symptoms of pregnancy and has been found to be equivalent to a structured interview in determining prevalence of depression. Scores range from 0-30 with higher scores signifying higher severity of depressive symptoms. A cut-off score of 10 on the EPDS will be used in this study to indicate moderate depressive symptoms.
Time Frame: Timepoint 0 (<19 weeks gestation) to Timepoint 3 (6 month well child visit)
Population: All participants completing data collection at respective timepoints.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 122 | 177
units on a scale
  Timepoint 0 | 13.042 (0.435) | 12.855 (0.362)
  Timepoint 1: number analyzed (Participants) | 73 | 95
  Timepoint 1 | 7.000 (0.560) | 7.776 (0.490)
  Timepoint 2: number analyzed (Participants) | 71 | 92
  Timepoint 2 | 6.119 (0.580) | 6.545 (0.506)
  Timepoint 3: number analyzed (Participants) | 68 | 86
  Timepoint 3 | 6.662 (0.576) | 6.818 (0.506)
Statistical Analysis 1: Comparison: Control vs Intervention; Null hypothesis: There was no significant difference in depressive symptoms across those 4 timepoints; Test type: Other; p < 0.001, two-way ANOVA
Statistical Analysis 2: Comparison: Control vs Intervention; Null hypothesis: There was no significant difference between the two groups in depressive symptoms at T0 baseline, as well as at time points 1, immediately following the intervention, 2, 6 weeks after the infants' birth, and 3, 6 months after the infants' birth; Test type: Other; p < 0.001, two-way ANOVA
Statistical Analysis 3: Comparison: Control vs Intervention; Null hypothesis: There was no statistically significant interaction between the intervention group and time; Test type: Other; p < 0.001, two-way ANOVA

5. Primary Outcome: Change Self-reported Stress at Timepoint 0 to Timepoint 3
Description: The Perceived Stress Scale (PSS) is a scale measuring stress will be administered at each of the in-person meetings. This scale is a standardized measure of global stress designed to elicit the degree to which respondents find their lives unpredictable, uncontrollable, and overloading (three central components of stress). The minimum score is 0 and the maximum score is 40. A higher score is correlated with a higher amount of stress. A score of 20 or greater is the high stress cut-off and will be used in this study.
Time Frame: Timepoint 0 (<19 weeks gestation) to Timepoint 3 (6 month well child visit)
Population: All participants completing data collection at respective timepoints.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 122 | 177
units on a scale
  Timepoint 0 | 21.857 (0.562) | 21.971 (0.468)
  Timepoint 1: number analyzed (Participants) | 73 | 95
  Timepoint 1 | 15.278 (0.723) | 15.596 (0.633)
  Timepoint 2: number analyzed (Participants) | 71 | 92
  Timepoint 2 | 12.448 (0.750) | 13.420 (0.654)
  Timepoint 3: number analyzed (Participants) | 68 | 86
  Timepoint 3 | 13.971 (0.744) | 14.193 (0.654)
Statistical Analysis 1: Comparison: Control vs Intervention; Null hypothesis: There was no significant difference in stress across those 4 time points; Test type: Other; p < 0.001, two-way ANOVA
Statistical Analysis 2: Comparison: Control vs Intervention; Null hypothesis: There was no significant difference between the two groups in stress, as measured by the GAD-7, at T0 baseline, as well as at timepoint 1 (immediately following the intervention), timepoint 2 (6 weeks after the infants' birth) and timepoint 3 (6 months after the infants' birth); Test type: Other; p < 0.001, two-way ANOVA
Statistical Analysis 3: Comparison: Control vs Intervention; Null hypothesis: There was no statistically significant interaction between the intervention group and time; Test type: Other; p < 0.001, two-way ANOVA

6. Secondary Outcome: Birth Weight
Description: record of birth weight as recorded in patient's medical file
Time Frame: T2= 6-8 week postpartum visit
Population: Infant weight was not available for all participants who completed timepoint (i.e. delivered at outside institution)
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Control | Intervention
Number analyzed (Participants) | 68 | 82
grams | 3139.9 (740.3) | 3310.1 (732.6)

7. Secondary Outcome: Breastfeeding Initiation
Description: Initiation of breastfeeding according to self-report at Timepoint 2: "Did you ever breastfeed or try to breastfeed your baby?". Responses below indicated number of participants that responded "yes" to this question.
Time Frame: T2= 6-8 week postpartum visit
Population: Number of participants that completed Timepoint 2
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 71 | 92
Participants | 64 | 83

8. Secondary Outcome: Breastfeeding Duration
Description: Self-reported maintenance of breastfeeding at approximately 6 months postpartum, inclusive of participants that responded both breastfeeding only and combined breast and bottle feeding (formula vs breastmilk not specified in question to participants).
Time Frame: T3 = at 6 month well baby visit
Population: Number of participants who completed Timepoint 3
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 68 | 86
Participants | 18 | 34

9. Secondary Outcome: Mode of Delivery
Description: (C/S, Vaginal, Forceps/Vacuum)
Time Frame: T2= 6-8 week postpartum visit
Population: Delivery mode not available for all participants who completed timepoint (i.e. delivered at outside institution)
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 69 | 85
Participants
  Vaginal Delivery | 52 | 52
  Assisted Vaginal Delivery (forceps, vacuum) | 0 | 4
  Cesarean Delivery | 17 | 29

10. Secondary Outcome: Nutritional Intake
Description: Nutrition behaviors as reflected in response to likert scale-type question "I eat fresh fruits and vegetable snacks". Reponses included Strongly Disagree (1), Disagree (2), Neither Agree Nor Disagree (3), Agree (4), Strongly Agree (5).
Time Frame: Timepoint 0 (<19 weeks gestation), T1 = 31 gestational weeks, T2= 6-8 week postpartum visit, T3 = at 6 month well baby visit
Population: Each row represents a study timepoint. Number analyzed in the number of participants who completed the respective timepoint.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 122 | 177
units on a scale
  Timepoint 0 | 3.955 (0.088) | 4.070 (0.073)
  Timepoint 1: number analyzed (Participants) | 73 | 95
  Timepoint 1 | 4.264 (0.098) | 4.298 (0.085)
  Timepoint 2: number analyzed (Participants) | 71 | 92
  Timepoint 2 | 4.075 (0.101) | 4.200 (0.090)
  Timepoint 3: number analyzed (Participants) | 68 | 86
  Timepoint 3 | 4.169 (0.103) | 4.173 (0.092)

11. Secondary Outcome: Level of Exercise
Description: Fitbit Flex 2 Accelerometer report data: data from Fitbit Flex 2 report will be collected at each of the in-person meetings
Time Frame: T1 = 31 gestational weeks, T2= 6-8 week postpartum visit, T3 = at 6 month well baby visit
Population: Fitbit data was not analyzed. Prior to COVID-19, participant adherence to Fitbit use was low (reported difficulty with charging, losing Fitbit, not bringing to study sessions). With the onset of the COVID-19 pandemic, participants were not able to bring Fitbits to in-person appointments to complete syncing.
Arm/Group | Control | Intervention
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Gestational Age at Birth
Description: Gestational age at birth will be collected as reported on patient's medical chart
Time Frame: T2= 6-8 week postpartum visit
Population: Gestational age was not available for all participants who completed timepoint (i.e. delivered at outside institution)
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Control | Intervention
Number analyzed (Participants) | 68 | 82
weeks | 39.0 (1.9) | 38.8 (1.8)

13. Secondary Outcome: Weight
Description: weight in pounds
Time Frame: Timepoint 0 (<19 weeks gestation)
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Control | Intervention
Number analyzed (Participants) | 122 | 177
pounds | 174.3 (47.2) | 171.0 (46.7)

14. Secondary Outcome: Participant Body Mass Index (BMI)
Description: derived calculation from weight and height values reported at each of the in person meetings
Time Frame: Timepoint 0 (Baseline at screening), T1 = 31 gestational weeks, T2= 6-8 week postpartum visit, T3 = at 6 month well baby visit
Population: Number analyzed in each row reflects the number completed at respective timepoints. This data is missing due to remote data collection lacking weight measurement devices (COVID-19).
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Control | Intervention
Number analyzed (Participants) | 122 | 177
kg/m^2
  Timepoint 0 | 29.4 (7.6) | 29.2 (7.5)
  Timepoint 1: number analyzed (Participants) | 66 | 91
  Timepoint 1 | 33.1 (7.8) | 31.8 (7.9)
  Timepoint 2: number analyzed (Participants) | 58 | 83
  Timepoint 2 | 31.2 (7.3) | 29.7 (7.2)
  Timepoint 3: number analyzed (Participants) | 61 | 78
  Timepoint 3 | 31.0 (8.0) | 30.4 (8.0)

15. Secondary Outcome: Participant Height
Description: height in feet and inches will be recorded at each of the in person meetings
Time Frame: Timepoint 0 (Baseline at screening)
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Control | Intervention
Number analyzed (Participants) | 122 | 177
inches | 63.9 (3.0) | 63.9 (3.0)

16. Secondary Outcome: Group Prenatal Care Acceptability
Description: Survey addressing participant responses to prenatal care in a group setting with 12 Likert scale-type responses: strongly disagree, disagree, neutral, agree, and strongly agree. Participants were also provided a free text box.
  Reported are responses to the question "I would recommend group prenatal care to a friend".
Time Frame: T1=31 gestational weeks
Population: Number analyzed in the number that completed the group prenatal care acceptability form. This form was added 10/16/2019, after data collection had started.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 58 | 56
Participants
  Strongly Disagree | 0 | 0
  Disagree | 0 | 0
  Neutral | 1 | 0
  Agree | 15 | 16
  Strongly Agree | 42 | 40

17. Secondary Outcome: Program Evaluation: Delivery Method
Description: Separate forms for intervention and attention control that collected data regarding participant experience in study program as well as delivery method, virtually or in-person. Delivery method was ranked by participants 1-4 for preference: 1:1 in person, 1:1 by telehealth, in small group in person, in small group by telehealth.
Time Frame: Timepoint 3, approximately 6 months postpartum
Population: Participants who completed Timepoint 3 after June, 2021, when form was added. 1 participant in the control arm did not complete the question ranking prenatal care delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 31 | 31
Participants
  First choice 1:1 in person | 9 | 6
  First choice 1:1 by telehealth | 3 | 2
  First choice in small group in person | 9 | 17
  First choice in small group by telehealth | 9 | 6
  Missing data | 1 | 0

18. Secondary Outcome: COPE-P Acceptability
Description: Survey administered with likert-style scale exploring participant satisfaction with different aspects of COPE-P. Participant score range 1 (Strongly Disagree) - 5 (Strongly Agree). Minimum score of 21, maximum of 105. High scores indicate higher satisfaction with the COPE-P program and its elements.
Time Frame: Timepoint 2 (6 to 8 weeks postpartum)
Population: Intervention participants who completed COPE-P acceptability at Timepoint 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 86
score on a scale | 94.05 (9.06)

19. Secondary Outcome: Program Evaluation
Description: as for outcome 17
Time Frame: Timepoint 3, approximately 6 months postpartum
Population: Participants who completed Timepoint 3 after June, 2021, when form was added.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 31 | 31
Participants
  Program helpful: yes | 31 | 30
  Program helpful: no | 0 | 1

ADVERSE EVENTS:
Time Frame: From baseline (<19 weeks gestation) to collection of Timepoint 3, approximately 6 months postpartum.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/177
Serious Adverse Events (participants affected / at risk) | 0/122 | 3/177
Other Adverse Events (participants affected / at risk) | 6/122 | 6/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=122) | Intervention (N=177)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1) — Any attempt at self-harm by a participant
Fetal Demise (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) — Death of the fetus prior to delivery and after 20 weeks gestation
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Control (N=122) | Intervention (N=177)
Preterm Birth (Pregnancy, puerperium and perinatal conditions) | 6/71 (6) | 6/92 (6) — Delivery prior to 37 weeks gestation

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic impacted delivery of care requiring changes to methodology and impacting recruitment. Virtual sessions and timepoints were utilized, limiting data collection (e.g. measured weight vs participant report), the efficacy of Fitbit use (less frequent clinic visits resulted in less reminders to charge devices and lack of syncing at in-person sessions). Recruitment target was not met and attrition exceeded expectations leading to fewer participants analyzed than expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan: Ohio Study Protocol (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT03416010/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: New York Study Protocol (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT03416010/Prot_SAP_001.pdf
  • Informed Consent Form: Ohio Informed Consent Form (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT03416010/ICF_002.pdf
  • Informed Consent Form: New York Informed Consent Form (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT03416010/ICF_003.pdf